CLINICAL TRIAL: NCT02143791
Title: A Post-market Study Evaluating the Prodigy Neuromodulation System for the Management of Failed Back Surgery Syndrome or Chronic Intractable Pain of the Trunk and/or Limbs.
Brief Title: Evaluate St Jude Medical Prodigy Neuromodulation for FBSS or Chronic Pain of the Trunk and/or Limbs
Acronym: Prodigy-I
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NM-13-038-ID-SC
Record Dates: First submitted 2014-05-19; First posted 2014-05-21 (Estimated); Results first posted 2024-07-08 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-01

CONDITIONS: Chronic Pain
Keywords: SCS; Burst stimulation
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Burst and Tonic stimulation (Experimental): All subjects were required to receive BurstDR stimulation therapy for the first 3 months after permanent implant. Thereafter the stimulation mode could be changed to tonic stimulation depending on patient's preference or physician's discretion.
  Interventions: Procedure: Burst and Tonic stimulation

INTERVENTIONS:
Procedure: Burst and Tonic stimulation

SUMMARY:
The purpose of this study is to confirm long term efficacy and safety of the ProdigyTM neuromodulation system in the management of failed back surgery syndrome or chronic intractable pain of the trunk and/or limbs.

ELIGIBILITY:
Inclusion Criteria:

* Patient with chronic, intractable pain of the trunk and/or limbs, including unilateral or bilateral pain associated with the following: failed back surgery syndrome or intractable low back and/or leg pain
* Patient diagnosed with radiculopathy
* Patient diagnosed with neuropathic pain
* Patient is considered by the investigator as a candidate for implantation of a SCS system
* Patient is ≥ 18 years of age
* Patient must be willing and able to comply with study requirements
* Patient must indicate his/her understanding of the study and willingness to participate by signing an appropriate Informed Consent Form

Exclusion Criteria:

* Patient is diagnosed with ischemic pain
* Patient is diagnosed with arachnoiditis
* Patient is diagnosed with complex regional pain syndrome (CRPS I and II)
* Patient is diagnosed with peripheral vascular disease (PVD)
* Patient is diagnosed with diabetic neuropathic pain
* Patient is diagnosed with chronic migraine
* Patient is immune-compromised
* Patient has history of cancer requiring active treatment in the last 6 months
* Patient has a documented history of substance abuse (narcotics, alcohol, etc.) or substance dependency in the last 6 months
* Patients with a SCS system or implantable infusion pump implanted previously
* Patient has a life expectancy of less than one year
* Patient is pregnant or is planning to become pregnant during the duration of the investigation
* Patient is unable to comply with the follow up schedule
* Patient needing legally authorized representative
* Patient unable to read and write
* Patient is currently participating in another clinical investigation with an active treatment arm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2014-06; Primary Completion 2016-01 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tony Van Havenbergh, Principal Investigator — St Augustinus, Wilrijk, Belgium; Devyani Nanduri, Study Director — Abbott Medical Devices
Locations (21):
- Australia (3):
  - Metro Spinal Clinic, Caulfield
  - Frankston Pain Management, Frankston
  - Epworth Hospital, Richmond
- St Augustinus Ziekenhuis, Wilrijk, Antwerp, Belgium
- Germany (5):
  - Medizinische Einrichtungen der Universität zu Köln, Cologne
  - University Hospital, Düsseldorf
  - Hospital Gera, Gera
  - Universitätsklinik für Stereataktische Neurochirurgie, Magdeburg
  - Universitatsklinikum Tubingen, Tübingen
- St Vincents University Hospital, Dublin, Ireland
- Italy (3):
  - Azienda Ospedaliera Monaldi, Napoli
  - Az. Ospedaliero-Universitaria Pisana - Stabilimento Santa Chiara, Pisa
  - Az. Osp.S.Giovanni Addolorata, Roma
- Netherlands (3):
  - Medisch Spectrum Twente, Enschede
  - St Antonius Ziekenhuis, Nieuwegein
  - Stichting Alysis Zorggroep, Velp
- Hospital Virgen de Rocio, Seville, Spain
- University Hospital, Uppsala, Sweden
- United Kingdom (3):
  - Seacroft Hospital, Leeds
  - St Bartolomew's, London
  - James Cook University Hospital, Middlesbrough

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 126 subjects were enrolled, 1 discontinued the study prior to the baseline visit.
Groups:
- Observational Cohort: All enrolled patients.
Period: Enrolled
Arm/Group | Observational Cohort
Started | 125
Completed | 121
Not Completed | 4
Not completed — Withdrawal by Subject | 4
Period: Trial Stimulation
Arm/Group | Observational Cohort
Started | 121
Completed | 100
Not Completed | 21
Not completed — Lack of Efficacy | 21
Period: Burst Stimulation Only (3 Months)
Arm/Group | Observational Cohort
Started | 100
Completed | 92
Not Completed | 8
Not completed — Withdrawal by Subject | 4
Not completed — Missing Data | 4
Period: Any Programming (3-6 Months)
Arm/Group | Observational Cohort
Started | 92
Completed | 88
Not Completed | 4
Not completed — Withdrawal by Subject | 3
Not completed — Missing Data | 1
Period: Any Program (6-12 Months)
Arm/Group | Observational Cohort
Started | 88
Completed | 86
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Observational Cohort
Number analyzed (Participants) | 125
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70
  Male | 55
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Germany | 47
  Italy | 20
  United Kingdom | 20
  Belgium | 8
  Australia | 13
  Netherlands | 10
  Sweden | 4
  Spain | 3
Primary Diagnosis [Count of Participants; unit: Participants]
  Radiculopathy | 13
  Failed Back Surgery Syndrome (FBSS) | 98
  Other Pain Conditions | 14
Work Status [Count of Participants; unit: Participants]
  Full-time | 17
  Part-time | 18
  Not Working | 90
Did Subject's Pain Cause Subject to Stop Working [Count of Participants; unit: Participants] — Population: Only subjects who reported "Not Working" when asked about work status (N=90) answered this question.
  Participants
    number analyzed (Participants) | 90
    Yes | 58
    No | 25
    Not applicable | 7

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change From Baseline in Overall VAS at 3 Months
Description: Percentage change in pain relief at the 3- month follow-up visit compared to baseline visit, as measured by the Visual Analog Scale (VAS). The VAS scale with a 10 cm (or 100 mm) line to indicate pain intensity progression with no pain (0) on the left end and worst pain (100) on the right end. Percent change is calculated as "[(post baseline baseline)/baseline] *100%" with positive numbers to represent increases and negative numbers to represent decreases.
Time Frame: 3 months
Population: 92 patients completed 3 months, but 86 patients had Burst programs only and had available data for Baseline and the 3-month follow-up visit.
Measure: Mean (Standard Deviation); unit: Percentage change
Groups:
- Burst Patients With Available Data: Subjects reporting percentage of Pain relief as mentioned with VAS in the Prodigy I study.
Arm/Group | Burst Patients With Available Data
Number analyzed (Participants) | 86
Percentage change | -51.3 (36.1)

2. Secondary Outcome: Pain Relief
Description: Patient reported pain relief. Patients were asked to evaluate their pain relief over the past week in percentage with 0% being no pain relief and 100% being complete pain relief.
Time Frame: 3 Months
Measure: Mean (Standard Deviation); unit: percentage of pain relief
Groups:
- Burst/Tonic Stimulation: All subjects with Burst/Tonic stimulation available at the respective study visit were included
Arm/Group | Burst/Tonic Stimulation
Number analyzed (Participants) | 90
percentage of pain relief | 53.9 (28.5)

3. Secondary Outcome: Pain Relief
Description: as for outcome 2
Time Frame: 6 Months
Measure: Mean (Standard Deviation); unit: percentage of pain relief
Arm/Group | Burst/Tonic Stimulation
Number analyzed (Participants) | 84
percentage of pain relief | 56.4 (28.8)

4. Secondary Outcome: Pain Relief
Description: Patient reported pain relief. Patients were asked to evaluate their pain relief over the past week in percentage with 0% being no pain and 100% being complete pain relief.
Time Frame: 12 Months
Measure: Mean (Standard Deviation); unit: percentage of pain relief
Arm/Group | Burst/Tonic Stimulation
Number analyzed (Participants) | 86
percentage of pain relief | 55.5 (31.2)

5. Secondary Outcome: Change in Pain Catastrophizing Scale
Description: The pain catastrophizing scale (PCS) is a validated scale containing 13 items to assess thoughts and feelings about pain while a person is experiencing pain. The total of all 13 items results in a minimum of 0 and a maximum of 54; scores above 30 indicate clinically significant pain catastrophizing. The mean change was calculated based on the value at 12 months minus the value at baseline.
Time Frame: 12 Months
Population: 84 patients had available data at baseline and 12 months for pain catastrophizing
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Burst/Tonic Stimulation
Number analyzed (Participants) | 84
score on a scale | -13 (15)

6. Secondary Outcome: Number of Participants With Analgesic Reduction
Description: Patient reported analgesic usage during the 4 weeks preceding the 12-month follow-up visit, compared to the baseline visit. The amount of patients who decreased the dose are reported.
Time Frame: 12 Months
Population: 19 patients had data available for analgesic usage at baseline and 12 Months.
Measure: Count of Participants; unit: Participants
Arm/Group | Burst/Tonic Stimulation
Number analyzed (Participants) | 19
Participants | 3

7. Secondary Outcome: Change in Quality of Life
Description: Subjects were provided with the Euroqol-5 dimensions (EQ-5D) questionnaire at baseline and 12 Months follow-up visit. In that questionnaire, subjects were asked to indicate a score for their health on a scale where 100 would mean 'the best state he/she can imagine' and 0 would be the 'worst state he/she can imagine).
Time Frame: Baseline and 12 Months
Population: 125 subjects had available data for the EQ-5D questionnaire at baseline and 85 at the 12 Months follow-up visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Burst/Tonic Stimulation
Number analyzed (Participants) | 125
units on a scale
  Baseline | 46 (22)
  12 Months: number analyzed (Participants) | 85
  12 Months | 62 (23)

8. Secondary Outcome: Rate of Serious Adverse Events and/or Procedure/Device-related Adverse Events
Description: Adverse device effects were defined as adverse events related to the study procedures or the device. Serious events were those that resulted in-patient or prolonged hospitalization or were life-threatening.
Time Frame: from enrollment to 12 months follow up
Population: All enrolled subjects who were at risk for SAE's and ADE's
Measure: Number; unit: events
Arm/Group | Observational Cohort
Number analyzed (Participants) | 125
events
  Serious Adverse Events | 57
  Adverse Device Effects | 24

9. Secondary Outcome: Paresthesia Mapping at 3 Months Compared to the Empower Study
Description: Paresthesia mapping is expressed in percent of paresthesia areas as indicated by the patient on a gender specific body diagram. 87 subjects with Burst stimulation at 3 Months (Prodigy-I) were compared to 134 subjects with tonic stimulation at 3 Months (Empower).
Time Frame: 3 Months
Population: 92 patients completed 3 months, but 87 patients had Burst programs only and had available data for Baseline and the 3-month follow-up visit
Measure: Mean (Standard Deviation); unit: percentage of paresthesias
Groups:
- Subjects From Prodigy I Study: Subjects using Burst only at 3 Months with available data for paresthesia mapping.
Arm/Group | Subjects From Prodigy I Study
Number analyzed (Participants) | 87
percentage of paresthesias | 18.2 (10.6)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Observational Cohort
All-Cause Mortality (participants affected / at risk) | 0/126
Serious Adverse Events (participants affected / at risk) | 39/126
Other Adverse Events (participants affected / at risk) | 31/126
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Observational Cohort (N=126)
Coronary artery disease (Cardiac disorders) | 1 (1) — Need to implant a stent, coronary artery disease
acute cardiac decompensation (Cardiac disorders) | 1 (1)
cardiac catherization (Cardiac disorders) | 1 (1)
hypothyriodism (Endocrine disorders) | 1 (1)
Diverticulosis (Gastrointestinal disorders) | 1 (1) — Laparascopic sigmoid resection due to diverticulosis
upper abdominal pain (Gastrointestinal disorders) | 1 (1) — acute pancreatitis
Lead Breakage/Fracture (General disorders) | 1 (1) — lead breakage due to patients anatomical structure of the spine
Lead contacts mostly invalid (General disorders) | 1 (1)
Lead migration (General disorders) | 2 (2)
Pain medication intolerance (General disorders) | 1 (1)
Persistant pain and/or numbness IPG site only (General disorders) | 1 (1) — skinny patient, IPG sat uncomfortably in her abdominal region
Undesirable changes in paresthesia (General disorders) | 1 (1)
device uncomfortable (General disorders) | 1 (1) — device not implanted deep enough
opiate withdrawal (General disorders) | 1 (1)
Ear infection (Infections and infestations) | 1 (1)
Infection: IPG & Lead site (Infections and infestations) | 2 (2)
Infection: IPG site only (Infections and infestations) | 1 (1)
Infection: Lead site only (Infections and infestations) | 1 (1)
Infection: extension site only (Infections and infestations) | 1 (1)
CSF leakage (Injury, poisoning and procedural complications) | 1 (1)
malignant tumor (Investigations) | 1 (1) — need MRI for diagnose cancer
Fall (Musculoskeletal and connective tissue disorders) | 1 (1)
ISG arthrose (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in hip (Musculoskeletal and connective tissue disorders) | 1 (2)
Persistant pain and/or numbness: undetermined (Musculoskeletal and connective tissue disorders) | 1 (1)
iliosacral joint osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
pain in leg (Musculoskeletal and connective tissue disorders) | 1 (2)
pain in vertrebral region due to fall (Musculoskeletal and connective tissue disorders) | 1 (1)
Bladder cancer diagnosed (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Bladder cancer diagnosed
malignant tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
ataxic gait disturbance (Nervous system disorders) | 1 (1)
IPG migration (Product Issues) | 1 (1)
Lead breakage/fracture (Product Issues) | 2 (2)
Lead migration (Product Issues) | 3 (3)
Persistant pain and/or numbness: Lead site only (Product Issues) | 1 (1)
Undesirable changes in pain (Product Issues) | 2 (2)
bad connection IPG-extension (Product Issues) | 1 (1)
bad connection between lead and IPG (Product Issues) | 1 (1)
insufficient paresthesia coverage (Product Issues) | 1 (1)
Anxiety disorder (Psychiatric disorders) | 1 (1)
Inability to control urination (Renal and urinary disorders) | 1 (1)
ovarian abcess (Reproductive system and breast disorders) | 1 (1)
Pain at IPG pocket (Skin and subcutaneous tissue disorders) | 1 (1) — normal post implant fat necrosis over IPG
microcirculation disturbance right foot (Vascular disorders) | 1 (1)
peripheral artery disease (Vascular disorders) | 1 (1)
varicose vein surgery (Vascular disorders) | 1 (1)
varicose veins (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Observational Cohort (N=126)
Diarrhea and vomitting (Gastrointestinal disorders) | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 1 (1)
Undesirable changes in pain (General disorders) | 1 (1)
Opiate withdrawal (General disorders) | 1 (1)
Undesirable changes in paraesthesia (General disorders) | 3 (3)
Dental abcess (Infections and infestations) | 1 (1)
Infection: IPG site only (Infections and infestations) | 1 (1)
Infection: Lead site only (Infections and infestations) | 1 (1)
Respiratory infection (Infections and infestations) | 3 (3)
Urinary tract infection (Infections and infestations) | 1 (1)
Fall (Musculoskeletal and connective tissue disorders) | 3 (4)
Joint pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Knee effusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Unintended stimulation effects: muscle spasms or cramping (Musculoskeletal and connective tissue disorders) | 3 (3)
Related to bladder carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Headaches- post procedure (Nervous system disorders) | 1 (1)
High impedance (Product Issues) | 1 (1)
Lead breakage/fracture (Product Issues) | 2 (2)
Lead extension retraction (Product Issues) | 1 (1)
Lead migration (Product Issues) | 1 (1)
Persistent pain and/or numbness: undetermined (Product Issues) | 1 (1)
Undesirable changes in pain (Product Issues) | 2 (2)
Undesirable changes in paraesthesia (Product Issues) | 2 (2)
Undesirable changes in stimulation (Product Issues) | 2 (2)
Burning sensation at IPG site (Skin and subcutaneous tissue disorders) | 1 (1)
Subcutaneous tissue changes at implant site (Skin and subcutaneous tissue disorders) | 1 (1)
Wound site complication (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No